CLINICAL TRIAL: NCT00194350
Title: Evaluation of the Role of Factor V Leiden Mutation in Implantation Failure
Brief Title: Factor V Leiden Mutation and Implantation Failure
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Kurt T Barnhart, MD, MSCE, University of Pennsylvania
Other Study IDs: 704111
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Infertility
Keywords: Infertility; Factor V Leiden
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Test for Factor V Leiden gene mutation

SUMMARY:
The purpose of this study is to determine whether inherited thrombophilias (tendency toward blood clotting) increase the risk of failure of the embryo to implant in IVF. The specific condition to be studied is the presence or absence of the Leiden mutation of the Factor V gene.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing in-vitro fertilization with successful ovarian hyperstimulation, oocyte retrieval, and fertilization
* Transfer of at least 2 fresh embryos of Grade 2 (preembryo with blastomeres of equal size and <=10% cytoplasmic fragmentation) or better

Exclusion Criteria:

* Infertility due to uterine anatomic defect
* Current use of anticoagulant medication, such as heparin or aspirin
* Known presence of any other condition associated with increased risk of thrombosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing in-vitro fertilization with successful ovarian hyperstimulation, oocyte retrieval, and fertilization; and the transfer of at least 2 fresh embryos of Grade 2 (preembryo with blastomeres of equal size and <=10% cytoplasmic fragmentation) or better
Sampling Method: Non-Probability Sample
Enrollment: 399
Dates: Start 2001-09; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania, United States